CLINICAL TRIAL: NCT04450290
Title: Dexamethasone-Eluting Cochlear Implant Electrode (CIDEXEL): A First in Human Study
Brief Title: Dexamethasone-Eluting Cochlear Implant Electrode
Acronym: CIDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MED-EL_CRD_2014_02
Record Dates: First submitted 2020-06-16; First posted 2020-06-29 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hearing Loss, Sensorineural; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: First-in-human, single-arm, exploratory, open-label, prospective, longitudinal, monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm - treatment (Experimental): All subjects will be implanted with the investigational device.
  Interventions: Device: CIDEXEL implant

INTERVENTIONS:
Device: CIDEXEL implant — The newly developed MED-EL Cochlear Implant incorporates the anti-inflammatory agent dexamethasone (DEX) into the electrode array. The passive elution of DEX during the post-implantation period has the purpose of counteracting the increase of the post-operative impedance induced by the insertion trauma.

SUMMARY:
A newly developed MED-EL Cochlear Implant incorporates the anti-inflammatory agent dexamethasone (DEX) into the electrode array. The passive elution of DEX during the post-implantation period has the purpose of counteracting the increase of the post-operative impedance induced by the insertion trauma.

The aim of this clinical investigation is to obtain a first experience in use of the investigational device in the adult clinical population, and to initially assess tools, techniques and performance outcome measures that may be considered in future clinical studies of similar devices.

DETAILED DESCRIPTION:
The principal objective of this study is to exploratively investigate the safety profile of the device which will be evaluated through the analysis of adverse events during the follow-up period. For the study to be considered a success, the results of the adverse event analysis shall never cause an unbalanced risk vs. benefit assessment.

The secondary objectives of this study aim at investigating the usefulness of possible outcome measures in evaluating the performance of the device.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of eighteen (18) years at time of enrolment.
* Severe to profound sensorineural hearing loss on the ipsilateral ear.
* A functional auditory nerve in the ear to be implanted.
* Subjects reporting to having used an optimally fit hearing aids for a minimum of three months before the decision that a cochlear implant (CI) is the preferential option.
* Cochlea anatomy compatible with the insertion of a +FLEX28 electrode array.
* Compatibility with a soft surgery approach as per clinical practice at the site.
* Post-lingual hearing impairment.
* Subject fulfilling indication criteria for a CI according to the local professional standards, as reported by the implanting surgeon.
* General health condition, psychological and emotional condition deemed compatible with the treatment and tests performed in this study and realistic expectations, as deemed appropriate by the implanting surgeon.
* Signed and dated informed consent before the start of any study-specific procedure.

Exclusion Criteria:

* Lack of compliance with any inclusion criterion.
* Previously having received a cochlear implant on the ear chosen for placing the IMD (Investigational Medical Device).
* Evidence of ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array or might cause increased risk of infection (e.g. dysplastic cochlea), as confirmed by medical examination and/or as per CT/MRT (Computed Tomography/Magnetic Resonance Tomography).
* Evidence of anatomic abnormalities that would prevent appropriate placement of the stimulator housing in the bone of the skull.
* Evidence of otosclerosis.
* Known allergic reaction or intolerance to the materials used in the implant (including medical grade silicone, platinum, iridium, parylene c, dexamethasone).
* Known absence of cochlear development or if the cause of deafness is non-functionality of the auditory nerve and/or the upper auditory pathway.
* Evidence of active external or middle ear infection or history of recurrent middle ear infection in the ear to be implanted.
* Evidence of perforated tympanic membrane in the ear to be implanted.
* Patient reporting immunosuppressive therapy or corticosteroids therapy in the 4 weeks before enrolment.
* Evidence of concomitant use of medicinal substances that, in the opinion of the investigator, could alter the therapeutic efficacy of dexamethasone.
* Unwillingness or inability of the candidate to comply with all investigational requirements.
* Evidence of medical contraindications to surgery of the middle and inner ear and anaesthesia.
* Additional disabilities that would prevent or restrict participation in the audiological and medical evaluations required of the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 10 months
  Safety profile of the device which will be evaluated through the analysis of adverse events

SECONDARY OUTCOMES:
IFT (Impedance Field Telemetry) - impedance | 10 months
  Impedance Field Telemetry and derived values
Electrically Evoked Compound Action Potential | 10 months
  Electrically Evoked Compound Action Potential and derived values
MCL (Maximum Comfortable Loudness) | 10 months
  Maximum Comfortable Loudness Levels and Thresholds
THR (Threshold) | 10 months
  Thresholds
PTA (Pure Tone Audiometry) Audiometrical values | 10 months
  Results from PTA assessment
Hearing Preservation rate | 10 months
  Rate of Hearing Preservation according to Skarżyński et al.
HSM (Hochmair-Schulz-Moser Sentence) Test | 10 months
  Speech test in noise
Questionnaire | 10 months
  Surgical feedback questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lenarz, Prof. Prof. h. c. Dr. med., Principal Investigator — Hals-Nasen-Ohrenklinik der Medizinischen Hochschule Hannover
Locations (1):
- MHH - Medizinische Hochschule Hannover, Hanover, Germany